CLINICAL TRIAL: NCT07073560
Title: Anthropometric Measurements Versus Radiologic Parameters of Hand Bones for Sex Identification in Upper Egypt Population: A Comparative Study.
Brief Title: Anthropometric Measurements Versus Radiologic Parameters of Hand Bones for Sex Identification
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aswan University (Other)
Responsible Party: Principal Investigator, Hadeer Mahmoud Mohamed Saleh, Demonstrator at forensic medicine and clinical toxicology, Faculty of medicine, Aswan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Human Sex Identification
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-04

CONDITIONS: Sex Determination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Males only (Active Comparator): About 60 of male participants and will be subjected to :
  1. Anthropometric hand measurements.
     -Left hands length, breadth and hand index will be estimated at first.
     -- The hand will be placed on a flat surface with the palm facing upwards and the fingers extended and close to each other.
  2. X-ray radiographs on the hand. The participants will undergo another examination by using 2D-images radiographs on the same hand. Posterior-anterior (PA) digital radiographs will be required for the left hand of the volunteers. The Osirix1 line-tool function will be used for measuring metacarpals on radiographs in (mm).
  Theses mrasurments:
  * Length superior ( LS )
  * Medullary length ( ML )
  * Mid-bone length ( MB )
  * Length of the base ( LB )
  Interventions: Procedure: Anthropometric Measurements
- Group B:Females only (Active Comparator): About 60 of female participants and will be subjected to :
  1. Anthropometric hand measurements.
     -Left hands length, breadth and hand index will be estimated at first.
     -- The hand will be placed on a flat surface with the palm facing upwards and the fingers extended and close to each other.
  2. X-ray radiographs on the hand. The participants will undergo another examination by using 2D-images radiographs on the same hand. Posterior-anterior (PA) digital radiographs will be required for the left hand of the volunteers. The Osirix1 line-tool function will be used for measuring metacarpals on radiographs in (mm).
  Theses mrasurments:
  * Length superior ( LS )
  * Medullary length ( ML )
  * Mid-bone length ( MB )
  * Length of the base ( LB )
  Interventions: Procedure: Anthropometric Measurements

INTERVENTIONS:
Procedure: Anthropometric Measurements — 1. Assessment of the accuracy of sex determination from hand indexes using anthropometric hand measurements.
  2. Assessment of the accuracy of sex determination from the length of the metacarpals using x-ray radiographs on the same hand.
  3. Determination of the best and least costly method for sex identification by comparing the effectiveness of the previous two methods.
  Other Names: Radiologic Measurements

SUMMARY:
Forensic anthropometry is the traditional and basic tool of forensic anthropology. It's the science of obtaining systemic measurements of the physical dimensions of the human body. This, in turn, is a very important parameter in personal identification.

Different anthropometric techniques are employed to determine sex from such fragmented body parts. Such anthropometric techniques aim to find cutoff points in the measurement of various body parts or bones that discriminate between males and females. Due to the effect of sex hormones, males are taller, larger and more strongly built than females, so measurements greater than the cutoff point are suggestive of a male and less than that are suggestive of a female.

DETAILED DESCRIPTION:
Personal identification is very challenging for forensic anthropologists.Various anthropological techniques can be used in identifying individuals. The 'big fours' of personal identification are determination of age, sex, stature and race. These form the features of 'tentative identification'.

Among these 'big fours' parameters , the determination of sex is not only considered one of the most important parameters; but it can primarily cut half of the possible number of matching identities.

But it is also one of the simplest tasks in forensic investigation if the whole body is available; as the external and internal genitalia directly suggest the sex; however, the problem arises when dismembered body parts are found.

Nowadays, there are increased events of murders where the mutilation of a dead body is done by murderer to destroy all traces of identity,and additionally, there are increased events of mass disasters where dismembered body parts are found.

The pelvis is the best sex-related body part indicator, with 95% accuracy. However, it may not always be available. Recent studies have worked towards the sex determination potentials of other body parts.

Hands are one of the most sexually dimorphic parts of the human body.Therefore, sex determination based on radiologic examination of hand bones and hand dimension anthropometric measurements is of considerable importance.

Since the use of image processing techniques (e.g., radiography and computed tomography) in sex determination by osteometric measurements of hand bones is costly.

ELIGIBILITY:
Inclusion Criteria:

* Egyptian volunteers of either sex who is above 18 years old and below 50 years old

Exclusion Criteria:

* Volunteers less than 18 years old or more than 50 years old.
* Volunteers with any of the following conditions will be excluded from this study as:
* Presence of any physical deformity, injury, fracture, or amputation in his/her hands.
* History of any surgical procedures involving the hands.
* Radiographs that show skeletal trauma or anomalies in the metacarpals.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Sex Determination | 6 months
  Evaluation of both males and females whom participated in the study for sex determination by comparing the accuracy of anthropometric hand measurements versus radiologic anthropometric parameters of hand bones

CONTACTS AND LOCATIONS:
Overall Officials: Randa Hussein Abdel Hady Mohamed, Professor, Study Chair — forensic medicine and clinical toxicology, Assuit Faculty of Medicine
Locations (1):
- Faculty of Medicine , Aswan University, Aswān, Egypt

IPD SHARING:
Plan to Share IPD: Undecided